CLINICAL TRIAL: NCT05528692
Title: The Time-Dependent Development of Incisional Hernias in Emergency Laparotomy Incisions of High-Risk Patients: a Danish Prospective Single-center, Non-randomized, Non-interventional, Observational Study
Brief Title: The Time-Dependent Development of Incisional Hernias in Emergency Laparotomy Incisions of High-Risk Patients
Acronym: MAGELA
Status: Withdrawn | Type: Observational
Why Stopped: Collaboration stopped
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Madeline Kvist, Principal Investigator, Herlev Hospital
Other Study IDs: HerlevH2
Record Dates: First submitted 2022-09-02; First posted 2022-09-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-11

CONDITIONS: Incisional Hernia; Emergency Midline Laparotomy
MeSH Terms: conditions — Incisional Hernia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging (MRI) — MRI is a non-invasive imaging modality capable of producing precise soft-tissue images in all body areas. In contrast to CT scanning, MRI does not rely on ionizing radiation. There are no known risks associated with MRI as long as patients with contraindications such as pacemakers are identified and excluded. The MRI scans in this study will be performed without use of contrast media.

SUMMARY:
The aim of this study is to describe the development of symptomatic and asymptomatic incisional hernias after emergency midline laparotomy over time in high-risk patients evaluated by consecutive MRI-scans.

DETAILED DESCRIPTION:
All patients operated with an emergency midline laparotomy in our clinic are potential participants and will be screened for participation. Potential participants will be briefly informed about the project by the hospital staff. If the patients are interested, they will be thoroughly informed about the study and asked to participate by one of the trial investigators before discharge.

Data will be obtained from the participants hospital files and by patient survey/interview. All data will be entered into a database using RedCap by trial investigators or their delegates.

Enrolled patients will be followed for two years. The trial involves four consecutive MRI-scans one month, three months, six months and two years after surgery. Change in quality of life, physical functioning and pain-score are also obtained by patient survey/interview at each visit. A concluding physical examination and abdominal wall ultrasound examination will be performed two years after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Unscheduled midline laparotomy in an emergency or subacute setting, involving perforated bowel, bowel obstruction, bowel ischemia (due to mesenteric vascular disease or incarceration), inflammatory diseases (e.g. diverticulitis, appendicitis, ulcerative colitis, cholecystitis and Crohn's disease), abscesses, non-traumatic intraabdominal bleeding or any emergency re-operation to elective surgery
* Age of 18 years or above
* BMI above 27
* At least one risk factor for incisional hernia i.e. earlier midline laparotomy, BMI > 30, abdominal aortic aneurysm or prior surgery for abdominal aortic aneurysm, active smoking, liver cirrhosis, re-laparotomy, age > 75, history of primary ventral hernia (treated or untreated before index surgery), large laparotomy involving more than 2/3 of the abdominal wall as measured from the xiphoid process to the pubic bone

Exclusion Criteria:

* Malign, incurable disease
* Other reasons for short life expectancy <2 year as evaluated by the investigator
* Midline-incisions <15 cm
* Mesh augmentation of abdominal wall closure at index surgery or earlier mesh augmentation of the abdominal wall
* Severe claustrophobia or any other mental habitus, making it impossible to perform MRI-scan without sedation
* Metallic magnetic implants that serves as a contraindication for MRI-scan (including pacemakers, large tattoos, insulin pumps, etc.)
* Metallic prosthetic non-magnetic implants that are suspected to create severe artefacts on the MRI-scan of the abdominal wall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient operated with an emergency midline laparotomy in our clinic will be evaluated for enrollment. Patients will be eligible if they comply with the listed inclusion and exclusion criteria.
  We aim to enroll 100 patients to ensure that 50 patients fulfill the study protocol. This is based on a risk of incisional hernia development of at least 30% over two years among the included high-risk participants, a two-year mortality of the participants as a group of 30% and a 20% loss to follow-up amongst the survivors.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Early (30-days) MRI-diagnosed, incisional hernia development in high-risk patients after emergency midline laparotomy. | 2 years

SECONDARY OUTCOMES:
MRI-diagnosed incisional hernia rates 3 months, 6 months and 2 years after laparotomy. | 2 years
Change in quality of life, physical functioning, clinical investigation and pain-score at 1 month, 3 months, 6 months and 2 years after laparotomy. | 2 years
Rate of MRI-verified subclinical vs. clinical detectable incisional hernias. | 2 years
30-day, 90-day, and 1-year mortality. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal- and Hepatic diseases, Surgical Section,, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All results, both positive, negative and inconclusive, will be attempted to be published in international English journals with external reviewers. Alternatively, the results will be published in another way.
Supporting Information: Study Protocol, ICF, CSR